CLINICAL TRIAL: NCT03920475
Title: An Investigation of the Role of Inflammatory Processes in the Development and Treatment of Idiopathic Unipolar and Bipolar Depression in Patients With Moderate to Severe Depressive Symptoms.
Brief Title: The Role of Inflammatory Processes in Development and Treatment of Depression
Acronym: INFLAME-D
Status: Completed | Type: Observational
Sponsor: Kliniken Essen-Mitte (Other)
Collaborators: University of Bordeaux (Other); IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other); Ruhr University of Bochum (Other); National Research Agency, France (Other); Créteil Hospital (Other); German Federal Ministry of Education and Research (Other Government); Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: EssenMitte
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Depressive Disorder; Depression; Inflammation
MeSH Terms: conditions — Depressive Disorder; Depression; Inflammation | interventions — Sertraline; Venlafaxine Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, edta, RNA-pax tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAU (treatment as usual) group: Patients with depression, meeting inclusion criteria, who needed antidepressant treatment and received either sertraline or venlafaxine.
  Interventions: Drug: Sertraline or venlafaxine; Diagnostic Test: Immune parameters

INTERVENTIONS:
Drug: Sertraline or venlafaxine — Patients were treated as needed with sertraline or venlafaxine following the official guidelines, starting with a dose of 25 mg/d or respectively 37,5 mg/day. The starting dose could be increased during the course of the treatment as clinically needed according to guide lines.
Diagnostic Test: Immune parameters — Serum was taken before, during an after treatment for measurement of different immune parameters.

SUMMARY:
The study investigates the influence of inflammatory processes on the development and the course of uni- and bipolar depression. It is assumed, that the concentrations of certain inflammatory proteins have an influence on the development of depression, its clinical severity, the response to treatment and the risk of relapse. To verify this hypothesis, a total of 145 patients, which were hospitalized für treatment of a depressive disorder in the study centers in Germany, Italy and France, were screened according to the criteria set out in the study protocol. Finally, 104 patients with moderate to severe depressive symptoms were included in the study. These patients were treated according to the recommendations of the DGPPN treatment guidelines. All patients received a medication with sertraline or venlafaxine during the study, starting at baseline. The patients were examined for the presence and severity of depressive symptoms at the time of study enrollment, as well as after 4 and 8 weeks, using standardized clinical test procedures. In addition blood was taken. In the serum of the patients, the concentrations of specific inflammatory proteins were measured using Cytometric Bead Array (CBA) and Enzyme-linked Immunosorbent Assay (ELISA) and then correlated with the clinical data. The investigated proteins include high-sensitivity CRP (C-Reactive-Protein), Interleukin 4, Interleukin 6, Interleukin 12, tumor necrosis factor-α, Eotaxin, Intercellular adhesion molecule 1 (CD54), Interferone-gamma and monocyte chemotactic protein 1 (MCP-1).

DETAILED DESCRIPTION:
The study investigates the influence of inflammatory processes on the development and the course of uni- and bipolar depression. It is assumed, that the concentrations of certain inflammatory proteins have an influence on the development of depression, its clinical severity, the response to treatment and the risk of relapse. To verify this hypothesis, a total of 145 patients, which were hospitalized für treatment of a depressive disorder in the study centers in Germany, Italy and France, were screened according to the criteria set out in the study protocol. Finally, 104 patients with moderate to severe depressive symptoms were included in the study. The severity of the symptoms was classified using well-established clinical rating scales like Montgomery-Asberg Depression Rating Scale (MADRS) and Hamilton rating scale for depression (HAMD). All enrolled patients were treated according to the recommendations of the German Association for Psychiatry, Psychotherapy and Psychosomatics (DGPPN) treatment guidelines.

In order to make drug-induced changes in the serum concentrations of the examined proteins as comparable as possible, it was determined in advance, that all patients should be treated with either sertraline (first choice) or venlafaxine (second choice) as an oral antidepressant. Apart from that, the antidepressive therapy, ie psychotherapy and similar procedures, had not been standardized. The treatment of study participants did not differ from the treatment of other patients hospitalized because of depression, who did not participate in the study. The patients were examined for the presence and severity of depressive symptoms at the time of study enrollment, as well as after 4 and 8 weeks, using standardized clinical test procedures. In addition blood was taken. In the serum of the patients, the concentrations of specific inflammatory proteins were measured using Cytometric Bead Array (CBA) and Enzyme-linked Immunosorbent Assay (ELISA) and then correlated with the clinical data. The investigated proteins include high-sensitivity CRP (C-Reactive-Protein), Interleukin 4, Interleukin 6, Interleukin 12, tumor necrosis factor-α, Eotaxin, Intercellular adhesion molecule 1 (CD54), Interferone-gamma and monocyte chemotactic protein 1 (MCP-1).

ELIGIBILITY:
Inclusion Criteria:

* Patients with uni- or bipolar depression, diagnosed according to the criteria of the Diagnostic and Statistical Manual Version IV (DSM-IV) via Mini-international neuropsychiatric interview Version 6.0 (MINI 6.0) diagnostic tool.
* At the time of inclusion in the study, the symptoms must meet at least the requirements of a moderately severe depression, defined by a minimum score of ≥ 22 on the Montgomery-Asberg Depression Scale.

Exclusion Criteria:

* Patients with severe somatic, rheumatic, endocrine or neurological comorbidities. This includes in particular neurological disorders associated with cognitive disorder, severe liver, kidney and cardiac diseases.
* Patients, who are being treated permanently with anti-inflammatory or immunosuppressive drugs (e.g. corticosteroids or alpha / beta-a(nta)gonists, immuno suppressant drugs).
* Patients with severe psychiatric disorders (Axis I) such as schizophrenia, dementia, attention deficit hyperactivity disorder, obsessive-compulsive disorder, current alcohol, drugs or drug addiction.
* Patients who have already been treated unsuccessfully with sertraline and all alternate medications allowed in the study.
* Pregnant or lactating (breast feeding) women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pharmacological treatment of depressive symptoms (out- or inpatient treatment).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Change in severity of depressive symptoms | 4 and 8 weeks after enrollment in the study
  Measurement of depressive symptoms using the Montgomery-Asberg Depression Rating Scale. The scale measures the severity of depression-associated symptoms. The usual cutoff points are 0 to 6 - depression absent, 7 to 19 - mild depression, 20 to 34 - moderate depression, >34 severe depression

SECONDARY OUTCOMES:
Changes in serum-concentration of inflammatory proteins | 4 and 8 weeks after enrollment in the stuy
  measurement of inflammatory proteins as listed in description of the study: high-sensitivity CRP (C-Reactive-Protein), Interleukin 4, Interleukin 6, Interleukin 12, tumor necrosis factor-α, Eotaxin, Intercellular adhesion molecule 1 (CD54), Interferone-gamma and monocyte chemotactic protein 1 (MCP-1). All results are given in the unit pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schäfer, Study Director — Kliniken Essen-Mitte

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) completely anonymized
Supporting Information: Study Protocol, ICF
Time Frame: starting 6 months after publication
Access Criteria: the data will be provided for the purpose of meta-analysis to scientific groups and researchers after personal request via the office of the studies director Prof. Martin Schäfer.